CLINICAL TRIAL: NCT01747590
Title: Imaging the Effects of Zolpidem and Alprazolam in Healthy Volunteers at 3T
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephanie C. Licata, Ph.D., Assistant Professor, Department of Psychiatry, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2011P000058; K01DA023659 (NIH)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Psychotropic Drugs Effects
MeSH Terms: interventions — Zolpidem; Alprazolam; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zolpidem, Alprazolam, Caffeine, and Placebo (Experimental): The 4 medications are given in a counterbalanced design.
  Interventions: Drug: Zolpidem; Drug: Alprazolam; Drug: Caffeine; Other: Placebo

INTERVENTIONS:
Drug: Zolpidem
  Other Names: Ambien
Drug: Alprazolam
  Other Names: Xanax
Drug: Caffeine
  Other Names: No Doz
Other: Placebo

SUMMARY:
The primary goal of this double-blind, placebo-controlled, within-subjects functional neuroimaging study is to examine the extent to which the hypnotic zolpidem decreases brain activity in regions of the brain known to process emotional information. Although zolpidem is an effective sleep-aid, its ability to engender anti-anxiety effects is equivocal, yet promising. Zolpidem's activity during tasks that engage anxiety-related processes in the brain will be compared to that of the known anxiolytic drug alprazolam, a positive comparator caffeine, and placebo. A secondary goal of this study is to compare the subjective drug effects, or how individuals feel, following the interventions. These measures will be used to determine the existence of brain-behavior relationships, thus demonstrating that imaging is an important tool for informing us about how drugs produce their effects in the brain.

DETAILED DESCRIPTION:
Benzodiazepines (BZs) and related drugs commonly are prescribed for treating anxiety and sleep disorders. Their clinical utility is based on their behavioral effects which are attributed to positive allosteric modulation of the GABA-A receptor. Multiple subtypes of the GABAA receptor exist, and recent research has focused on understanding the role of BZ-sensitive GABAA receptors (i.e., receptors containing alpha-1, alpha-2, alpha-3, and alpha-5 protein subunits) in the behavioral effects of BZ-type drugs. Results from a body of work suggests that the anxiolytic or anti-anxiety effects of BZ-like drugs likely involve alpha-2- and/or alpha-3-containing GABAA receptors, while their sedative-like effects are attributable to alpha-1GABAA receptors.

Compared to BZs, the BZ-like hypnotic zolpidem exhibits relative selectivity for alpha-1GABAA receptors. Although this selectivity is believed to underlie its superior hypnotic ability, zolpidem's ability to engender anxiolytic-like effects has been inconsistent. Zolpidem's primary effects should not include anxiolysis given its preference for interacting with alpha-1GABAA receptors and their abundant distribution in sensorimotor cortex and extrapyramidal motor areas relative to the more enriched distribution of the other receptor subtypes throughout the limbic system, anterior thalamus, and caudate nucleus. However, in the amygdala, a brain region that has been shown to be intricately involved in anxiety-related neuronal processes, high levels of alpha-1 GABAA receptors as well as alpha-2 and alpha-3GABAA receptors are expressed.

Among the anxiety-related processes typically studied empirically, the ability to recognize emotion is an important proxy for psychopathology. Neuroimaging studies have shown that the ability to process emotional stimuli requires coordinated activity between the amygdala, insula, and prefrontal cortical regions. Individuals who suffer from anxiety disorders exhibit an impaired ability to recognize facial emotion, which has been associated with aberrant amygdala activation. Importantly with respect to pharmacological manipulation of anxiety-related brain function, functional magnetic resonance imaging (fMRI) studies examining the neural correlates of emotional processing by employing acute challenge with potent anxiolytics have demonstrated significant reductions in the blood oxygen level-dependent (BOLD) signal within the amygdala and insula.

The primary aim of the study outlined in this protocol is to demonstrate drug-induced differences in limbic activation during an fMRI-based emotional face recognition task following acute administration of zolpidem, alprazolam, and the positive control caffeine in healthy volunteers. Although zolpidem may exhibit a similar behavioral pharmacological profile to the conventional BZs in many instances, its relative GABAA receptor selectivity distinguishes it from its non-selective counterparts. Thus it is hypothesized that the anxiolytic alprazolam (1 mg) will reduce the BOLD response to emotional faces within the amygdala and insula similar to other anxiolytics (e.g., lorazepam, diazepam, and pregabalin), while the hypnotic zolpidem (10 mg) will not cause such a reduction. It is hypothesized further that because adenosine receptors have been localized to the amygdala and caffeine has been shown to be anxiogenic, an acute challenge with a moderate dose of caffeine (200 mg) will enhance the BOLD response in the amygdala and/or insula during the face recognition task. The data that will be collected in this aim will provide the first in vivo brain imaging evidence for different actions based on the different GABAA receptor pharmacological profiles of zolpidem and alprazolam, and will support their clinical roles in the treatment of insomnia and anxiety, respectively.

The secondary aim of this project is to collect information regarding the subjective drug effects of each of the four interventions. This information, in conjunction with data showing how each treatment affects brain activity, permits the visualization of the neurobiological substrates of drug action. For instance, in a previous study we found that zolpidem-induced increases in self-reported ratings of "like", "high", and intoxication were related to increased brain activity in specific limbic networks. Our data were consistent with those areas shown previously to undergo hemodynamic or metabolic alterations in association with the subjective states of intoxication following administration of cocaine, alcohol, and hydromorphone, and they speak to a body of literature implicating limbic, paralimbic, and mesocortical regions in mediating the actions of psychotropic drugs. Because alprazolam is known to possess more abuse potential in general, results from the present study may confirm our previous findings while also demonstrating that investigating pharmacological effects on brain activity may help identify the neural correlates of drug action and behavior, thereby revealing the functional significance of GABAergic modulation on intrinsic brain activity.

A total of 12 healthy normal drug-naïve volunteers will be enrolled at McLean Hospital to participate in this 5-visit (1 screening visit, 4 study visits) double-blind, placebo-controlled study. Participants will be between 21 and 40 years of age, they can be either male or female, and there are no restrictions regarding ethnic background. Participants will have no past or current neurological or psychiatric disorders (including any substance abuse and/or dependence), no family history of alcoholism, no medical conditions that could affect drug disposition, and they will not be taking any medications. Participants also cannot have any MRI scanning contraindications (including pregnancy). They must be able to provide informed consent.

Volunteers will visit the laboratory for a screening visit during which s/he will sign the informed consent form, and undergo both physical and psychiatric exams. The second, third, fourth, and fifth visits will involve pre-study assessments, a standard breakfast, questionnaire sets, drug treatment, one scanning session, and lunch. After a baseline period during which participants will answer computerized questionnaires, they will receive a study medication (zolpidem [10 mg], alprazolam [1 mg], caffeine [200 mg], or placebo) and then answer the questionnaires. At 60-min post-medication, participants will be positioned within the scanner, and while in there they will perform tasks, blood pressure/heart rate will be monitored continuously, and an eye-tracking device will assess if their eyes are open. The scanning session will last approximately 1 hr, and it will be followed by hourly questionnaires sets until 6-hrs post-medication. Participants will take a taxicab home at that time. The entire visit will last approximately 8 hrs.

An exhaustive screening procedure ensures that participants entering the study have no contraindicating conditions. All procedures are performed by experts specifically trained in their respective areas to minimize risks, discomfort, and adverse events. Participants are well informed of the potential risks of the study. The informed consent form is detailed and explicit. Participants are provided with unlimited time to read the consent and study personnel review it in detail before participants sign. In addition, participants have the opportunity to ask questions before, during, and after consent and at any time during the study. Participants can earn up to a total of $500 for completing the study.

ELIGIBILITY:
* Participants will be right-handed male and female volunteers between the ages of 21-40
* Participants will consume between 100 and 300 mg caffeine on a daily basis
* Participants cannot meet DSM-IV criteria for lifetime and/or current mood, anxiety, psychotic, and alcohol/drug use disorders as identified by the SCID
* Participants must report ≤ 10 lifetime experiences with substances other than nicotine and alcohol
* Participants cannot be taking any prescription medication (except certain short-term anti fungal agents and some topical creams for dermal conditions)
* Participants cannot be taking any psychotropic medications
* Non-smoking participants are preferred, but will admit those who smoke less than 5 cigarettes per day
* Participants cannot have a history of major head trauma resulting in cognitive impairment, seizure, or other neurological disorders.
* Participants cannot have any conditions that are contraindicated for MRI
* Participants cannot have a family history of alcoholism
* Participants cannot have any abnormal blood chemistries/urinalysis results, current or past cardiac problems, or any other medical condition that may affect drug disposition (e.g., Hepatitis C)
* Participants cannot be taking oral contraceptives (Kalow and Tank, 1991; O'Connell, 1995) or be pregnant
* Participants must be able to read screening materials including consent form and give informed consent

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood oxygen level-dependent (BOLD) signal as measured with fMRI | 45 min after drug administration

SECONDARY OUTCOMES:
Change in subjective drug effects as measured by self-report questionnaires | Over the course of 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie C Licata, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States